CLINICAL TRIAL: NCT04674735
Title: Multicentre, Open Label, Phase I Clinical Trial to Evaluate the Safety of APSLXR for the Treatment of Vertigo of Vestibular Origin or Meniere's Disease
Brief Title: Safety of APSLXR in Patients Presenting Vertigo of Vestibular Origin or Meniere's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Cancelled by Sponsor
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APS004/2020
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Meniere Disease; Vertigo; Vertigo Vestibular
MeSH Terms: conditions — Meniere Disease; Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APSLXR (Experimental)
  Interventions: Drug: APSLXR

INTERVENTIONS:
Drug: APSLXR — Oral coated tablets once a day for 60 days.

SUMMARY:
The purpose of this study is to evaluate the safety of APSLXR in participants with Meniere's disease or other Verigo of vestibular origin. Pharmacokinetics will also be evaluated in a small group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Meniere's Disease or Vertigo of Vestibular Origin;
* Voluntarily consent to participate in the study;

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding;
* Participants presenting uncontroled systolic hipertension (>140/90 mmHg);
* Participants presenting uncontroled diabetes (blood glucose >200 mg/dL).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | during 60 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters in steady state | at Day 60
  Cmáx_SS

IPD SHARING:
Plan to Share IPD: No